CLINICAL TRIAL: NCT03435809
Title: Randomized Control Study on the Impact of a Pozzi Tenaculum Forceps Use on the Success Rate of Intrauterine Insemination (IUI)
Brief Title: Pozzi Forceps in Intrauterine Insemination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUdeQuebec
Record Dates: First submitted 2018-02-03; First posted 2018-02-19 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Infertility; Insemination
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pozzi for intrauterine insemination (Active Comparator): Treatment done with a pozzi tenaculum forceps
  Interventions: Procedure: Intrauterine insemination
- No Pozzi for intrauterine insemination (Active Comparator): Treatment done without a tenaculum forceps
  Interventions: Procedure: Intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination — Obligatory use of a Pozzi forceps tenaculum during intrauterine insemination

SUMMARY:
Many infertility and subfertility issues are treated nowadays with intrauterine inseminations. This is a minimally invasive technique that consists in placing sperm into a woman's uterus. Inseminations have only a fair success rate despite advances in technology ( 7 % per cycle). The goal of this study is to find an easy intervention that could help with success rate. Some studies are showing that the use of Pozzi tenaculum forceps might increase rates of pregnancy following intrauterine inseminations. In order to study the impact of this intervention, we are conducting a randomized controlled trial comparing the rate of term live births after IUI between patients who had their treatment done with a pozzi tenaculum forceps and those who had their treatment done without a tenaculum forceps.

DETAILED DESCRIPTION:
Once the initial investigations are done, an oral treatment is started on the first cycle if medically indicated.

At mid-cycle, patients undergo a transvaginal ultrasound looking for follicles' maturation. This ultrasound's goal is to detect ovulation and plan the IUI. If no follicle is detected, the transvaginal ultrasound is repeated later. If there is no luteinizing hormone (LH) peak detected upon ovulation urine test, there will be an ovulation induction with human chorionic gonadotropin (hCG) based depending on patient's age, number and size of detected follicles. Subcutaneous hCG or intramuscular hCG can be used. A cycle can be cancelled if there is no ovulation or if there is ovarian hyperstimulation.

During ovulation, semen analysis is performed, looking at sperm volume, sperm concentration and mobility. Then, semen is treated with a density gradient or with centrifugation. Isolated sperm are diluted in 0.5 to 1 mL of media and maintained in an incubator at a 37 º C temperature until insemination. The laboratory performs a second analysis on the washed semen in order to obtain the most accurate measures. If donor's semen is used, the andrology laboratory prepares the specimen and then processes with the semen analysis.

Patients are inseminated the day after a spontaneous LH peak or 24-36h after ovulation induction. For those who are randomized to the intervention group, a pozzi tenaculum forceps will be applied and clamped horizontally to the anterior cervical labrum with only a single click and mild traction will be applied in another to decrease the uterocervical angle. When no tenaculum is applied, motion will be mimicked without actual tissue prehension. Patients randomized to the control group will only have a tenaculum forceps applied in cases where the IUI is not feasible otherwise by the gynecologist. Indeed, it is sometimes necessary, when the cervical anatomy does not allow for easy pass of the catheter, for a pozzi tenaculum forceps to be used in order to insert the insemination catheter properly in the uterine cavity. In that case, tenaculum use will be recorded in the patient's file. No cervical insemination is allowed. Insemination is performed with flexible catheters and care is taken to avoid touching the uterine fundus with the catheter tip. There are multiple catheters available in the gynecology clinic, namely catheters The Curve (Cooper Surgical, Berlin), Shapeable IUI Catheter (Thomas Medical, Indianapolis) and Mini space (Laboratory C.C.D., Paris). After the intervention, patients are instructed to lie flat for 10 minutes after which they go home until next appointment.

Intercourse is allowed following IUI treatments. Patients are instructed to perform a urinary pregnancy test at home to weeks after the IUI, which will be provided to them. If the test is positive, patients are scheduled for a transvaginal ultrasound on week #7 of amenorrhea to confirm proper intrauterine pregnancy evolution. When pregnancy is confirmed, patients are referred to an physician for obstetrical follow-up.

In case of treatment failure, patients go on with ovulation induction or stimulation for the next cycle as previously prescribed by the gynecologist at mid-cycle ultrasound, if indicated. Dosages of ovarian stimulation medication may be modified, at physician's discretion, in order to optimize response to treatment according to the usual indications (ovarian hyperstimulation, side effects, poor response, etc.) Patients will be followed for 3 cycles and, if need be, can receive subsequent IUI treatments outside research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infertility :Defined as no pregnancy after one year of regular unprotected vaginal intercourse
* Infertility secondary to endometriosis, to a mild to moderate male factor, to an ovulatory dysfunction, an unexplained infertility or any other known medical indication for IUI.
* Intrauterine insemination with a partner's semen sample or a donor sample
* First IUI treatment or first treatment since last pregnancy
* Ovulation induction with letrozole medication
* Being able to speak and understand French

Exclusion Criteria:

* Bilateral tubal occlusion
* Active pelvic infection
* < 1 X 10^6 mobile sperm on semen analysis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Rate of live births | 10 months after positive pregnancy test
  Live born delivery resulting from an intrauterine insemination cycle

SECONDARY OUTCOMES:
Clinical rate of pregnancy (urinary or blood b-hcG) | At the end of 1 cycle (approximately 28 days)
  Positive urinary pregnancy test ou blood test (b-hcG)
Patients' global satisfaction assessed by questionnaire | 15 minutes after the intervention
  In regards of the treatment they received, yes/no questions Are you satisfied with the treatment you received? Do you think this treatment is an reasonable option of treatment?
Pain Level on visual analog scale | 15 minutes after the intervention
  Measure from 0-100 in mm, 100 being the highest pain level On a scale from 0-10 with intermediate values, 10 being the worst pain ever and 0 being no pain at all.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve Bergeron, MD, Principal Investigator — CHUL (CHUdeQuebec) - Département d'endocrinologie de la reproduction
Locations (1):
- CHUL Centre Mère Enfant Soleil - CHU de Quebec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dufour S, Viau M, Cote M, Lefebvre J, Maheux-Lacroix S, Bergeron ME. Impact of a Pozzi tenaculum forceps use on the success rate of intrauterine insemination (IUI) : protocol for a randomised control trial. BMJ Open. 2021 Mar 18;11(3):e043230. doi: 10.1136/bmjopen-2020-043230. PMID 33737427